CLINICAL TRIAL: NCT04693533
Title: Fremanezumab, Migraine and Sleep
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We could not recruit enough patients who fulfilled inclusion criteria and eventually gave up and terminated the study. The reason for not closing it is that we did have
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Rami Burstein, Professor of Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020P-001191
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Migraine Disorders; Sleep Disorder
MeSH Terms: conditions — Migraine Disorders; Sleep Wake Disorders | interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- treatment effect (Other): No 2 arms and only 1 intervention
  Interventions: Drug: Fremanezumab Prefilled Syringe [Ajovy]

INTERVENTIONS:
Drug: Fremanezumab Prefilled Syringe [Ajovy] — The treatment is 225 mg (dissolved in 1.5 ml saline) fremanezumab. Fremanezumab (Ajovy) is a month-long-acting anti-CGRP injection that patients are taught to self-administer at home.

SUMMARY:
The main goal of this study is to determine whether there is a relationship between fremanezumab's ability to prevent migraine and improved sleep quality in migraine patients (fremanezumab is a FDA-approved humanized CGRP monoclonal antibody for the treatment of migraine).

This is a within-person study design that examines treatment effects (changes) using high-resolution assessments. To complete the study, each participant will be observed using daily assessments of migraine and sleep outcomes before treatment (baseline: 0 to 30 days), and at 1, 2, and 3 months after treatment (injection 1: days 31-60, injection 2: days 61-90, injection 3: days 91-120). In essence, this creates an interrupted time-series design where repeated interventions are introduced at fixed intervals.

DETAILED DESCRIPTION:
The study involves 5 visits to the headache clinic:

In clinic visit 1 (day 0), subjects will learn about the study and if they agree to participate, will be consented and screened for eligibility. Those deemed to be eligible will be asked to fill a headache questionnaire and then taught how to fill at home a daily e-diary for sleep and a daily e-diary for headache.

In clinic visit 2 (day 30), subjects will return to the headache clinic to review their e-diaries and receive the first treatment. The treatment is 225 mg (dissolved in 1.5 ml solution) fremanezumab. Fremanezumab is a monthly dosed anti-CGRP mAb injection.

In clinic visit 3 (day 60), we will review participants' headache and sleep diaries 1 month after receiving the 1st injection and administer the 2nd injection. This appointment will be conducted by either one of the study physicians or the study nurse.

In clinic visit 4 (day 90), we will review participants' headache and sleep diaries 1 month after receiving the 2nd injection and and administer the 3rd injection. This appointment will be conducted by either one of the study physicians or the study nurse.

In clinic visit 5 (day 120), participants will return to the headache clinic to summarize their experience, review their 120-days e-diaries, and provide any feedback they may have about their experience with fremanezumab.

Assessments of headache and sleep:

At screening (visit 1), headache severity and impact will be assessed based on patients' interviews and HIT-6. Sleep quality will be assessed using the Insomnia Severity Index. (https://cbtscience.files.wordpress.com/2014/02/insomniaseverityindex.pdf).

On days 30, 60, 90 and 120, baseline and treatment impact on headache and sleep will be assessed using the Headache e-diary and the consensus sleep diary [Carney et al., (2012) The consensus sleep diary: Standardizing prospective sleep self-monitoring, Sleep Vol.35, No.2, pp.287-302], the latter of which captures total sleep time, sleep latency, wake after sleep onset, number of awakenings, quality, sleep efficiency, and trouble staying awake.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65 years
* Been previously diagnosed with migraine (with or without aura), in accordance with the ICHD-3 criteria
* Experiences between 10 to 25 headaches days per month (during the last 3 months), with at least 8 of them being migraine days during which the migraines lasted more than 4 hours if untreated
* Onset of migraine at age 50 years or younger
* Agrees to refrain from initiating or changing the type, dosage, or frequency of any prophylactic medications for indications other than migraine that may interfere with the study objectives (e.g., antidepressants, anticonvulsants, beta-adrenergic blockers, etc.)
* Able to provide written informed consent
* Scoring 10 or higher on the Insomnia Severity Index (8-14 = subthreshold insomnia, 15-21 = clinical insomnia of moderate severity, 22-28 = clinical insomnia of severe severity)

Exclusion Criteria:

* -
* Currently on a regimen of 1 or more migraine preventative therapy
* Other significant pain problem (e.g., cancer pain, fibromyalgia, other head or facial pain disorder) that may confound the study assessments
* Known or suspected severe cardiac disease (e.g., symptomatic coronary artery disease, prior myocardial infarction, congestive heart failure)
* Known or suspected cerebrovascular disease (e.g., prior stroke or transient ischemic attack, symptomatic carotid artery disease, prior carotid endarterectomy or other vascular neck surgery)
* Abnormal baseline electrocardiogram (ECG) within the last year (e.g., second or third-degree heart block, prolonged QT interval, atrial fibrillation, atrial flutter, history of ventricular tachycardia or ventricular fibrillation, clinically significant premature ventricular contraction)
* Uncontrolled high blood pressure (systolic >160 mm HG, diastolic >100 mm Hg) after 3 measurements within 24 hours
* Known history or suspicion of secondary headache
* Known history or suspicion of substance abuse or addiction (within the last 5 years)
* Currently using marijuana (including medical marijuana) or has used marijuana (including medical marijuana) or cannabidiol oil within the last 1 year
* Currently takes simple analgesics or NSAIDs >15 days per month or triptans, ergots, or combined analgesics >10 days per month for headaches or other body pain
* Currently takes prescription opioids for headaches or body pain
* Undergone nerve block (occipital or other) in the head or neck within the last 3 months
* Received botulinum toxin or anti-CGRP-mAb injections within the last 6 months
* Nursing, pregnant or thinking of becoming pregnant during the study period, or of childbearing years and unwilling to use an accepted form of birth control
* Participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days
* Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with the follow-up requirements, or provide self-assessments is compromised.
* A relative of or an employee of the Investigator or the clinical study site
* Psychiatric or cognitive disorder and/or behavioral problems that, in the opinion of the clinician, may interfere with the study
* History of claustrophobia
* Diagnosis of obstructive sleep apnea or restless legs syndrome
* BMI of 30 or greater
* Daily use of sleep-promoting drugs. These include eszopiclone; zaleplon; zolpidem; benzodiazepines (estazolam, flurazepam, quazepam, temazepam, triazolam); barbiturates (amobarbital, amobarbital-secobarbital, chloral hydrate); doxepin; quetiapine; ramelteon; trazodone; suvorexant; lemborexant; OTC nighttime meds (doxyalamine; diphenydrame); and melatonin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Fremanezumab and sleep | 4 months
  This primary outcome measures improvement in sleep quality during the treatment period as compared to the pre-treatment period. Sleep quality will be measured using the Insomnia Severity Index. This index scores requires subjects to answer 7 questions by depicting a number (between 0 and 4 ) that represents best their answer. The scale of the Insomnia Severity Index is 0-28. The total score categories are as follows: 0-7 = No clinically significant insomnia, 8-14 = Subthershold insomnia, 15-21 = Clinical insomnia (moderate severity), 22-28 = Clinical insomnia (severe).
Fremanezumab and migraine | 4 months
  This primary outcome measures changes in number of migraine days per month before and during treatment. The number of migraine days per month will be captures using a validated headache questionnaire and scores as follows: 0-8 migraine days per month = low frequency episodic migraine, 9-14 migraine days per month = high frequency episodic migraine, 15-30 migraine days per month = chronic migraine.

CONTACTS AND LOCATIONS:
Overall Officials: Sait Ashina, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC Headaceh Clinic, Boston, Massachusetts, United States